CLINICAL TRIAL: NCT02055625
Title: Treatment of Oral Mucosa in Patients With Graft-versus-host Disease Following Injection of Mesenchymal Stem Cells - Human Pilot Study
Brief Title: Mesenchymal Stem Cells as a Treatment for Oral Complications of Graft-versus-host Disease
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Rachael Sugars, Associate Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/1241-31/1
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Graft -Versus-host-disease
Keywords: Graft-versus-host-disease; Immune system diseases; Oral
MeSH Terms: conditions — Graft vs Host Disease; Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mesenchymal stromal cell treatment (Experimental): Biological: Mesenchymal stromal cells
  Interventions: Biological: Mesenchymal stromal cells

INTERVENTIONS:
Biological: Mesenchymal stromal cells — Allogenous mesenchymal stromal cells will be injected directly underneath the mucosal lesions at one side under local anesthetic at 2.5-4 million cells/ml. A total of approximately 1.7 ml will be injected divided in 2-3 injections around the lesion. Patients will be followed every second day up to 7 days afterwards and then routinely at 14 days, 1 month, 2 months and 6 months to assess the healing process.

SUMMARY:
Graft-versus-host disease (GVHD) is a major complication of allogeneic hematopoietic stem cell transplantation (HSCT), and is classified as acute (aGVHD) or chronic (cGVHD). aGVHD onsets within the first 100 days after transplant or with clinical features including erythema, liver dysfunction and oral mucositis, whilst cGVHD or persistent GVHD occurs in approximately 30-60% of transplant patients who survive their first year . Long-term five-year prognosis for cGVHD patients is poor with a 70% mortality rate. cGVHD manifests as an autoimmune-like disease affecting multiple sites, including skin, mouth, eyes, gastrointestinal tract, liver, and joints. The oral cavity is the second most common site to be affected with symptoms in 45-83% of cases. In the mouth a diverse spectrum of clinical features can be found for example mucosal lesions can affect almost any site, salivary gland dysfunction and restricted mouth opening. Short-term patients can experience mucosal sensitivity, malnutrition, problems speaking, increased caries risk, xerostomia, oral pain and a diminished quality-of-life. Long-term complications include secondary malignancies and perhaps early death. Clinical management seeks to alleviate the symptoms and improve quality-of-life but 50% of patients fail front-line systemic steroid therapy. Oral cGVHD can be treated with topical high potency corticosteroids and oral rinses, however these treatments are not always effective and carry a risk of systemic absorption. Mesenchymal stem/stromal cells (MSCs) resident in adult and fetal tissues, such as the bone marrow have the capacity to form bone, cartilage, stroma, muscle and fat, are known to exhibit immunosuppressive and immunoregulatory properties both in vivo and in vitro. MSC infusions have been used to treat disorders such as osteogenic imperfecta, cardiovascular disease and to heal large bony defects. Indeed, the immunosuppressive capacity of MSCs have led to infusions being used as a second-line treatment for GVHD patients, and our group has shown within a Phase II clinical trial, 55% aGVHD patients who failed front-line steroid treatment responded to MSC infusion these studies are going with cGVHD patients. The goal of this project is to perform a pilot study to determine whether MSC injections directly into mucosal lesions in patients with oral cGVHD are able to alleviate the symptoms and facilitate the reparative process.

ELIGIBILITY:
Inclusion Criteria:

* Chronic graft-versus-host disease and oral manifestations grade 3 exhibiting severe symptoms, according to the NIH Consensus Working Group for Diagnosis and Staging of cGVHD and have failed frontline therapy

Exclusion Criteria:

* Active malignancy
* Fulfilling criteria for previously initiated study for treatment of chronic graft-versus-host disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Change in disease activity according to National Institutes of Health criteria for oral graft-versus-host disease | Baseline to 6 months

SECONDARY OUTCOMES:
Change in self-assessed disease activity and quality of life | Baseline to 6 months
Safety | Baseline to 21 months
  Frequency of complications, infections and relapse

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Le Blanc, Professor, Principal Investigator — Karolinska Institutet; Karin Garming-Legert, DDS, PhD, Principal Investigator — Karolinska Institutet; Rachael Sugars, BSc, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Oral and Maxillofacial Surgery, Karolinska Univeristy Hospital, Stockholm, Huddinge, Sweden